CLINICAL TRIAL: NCT00718874
Title: Dietary Intervention to Improve Insulin Dynamics During the Pubertal Transition
Brief Title: A Specialized Diet for the Unique Metabolic Characteristics of Peripubertal African American Girls
Acronym: PRIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Krista Casazza, Krista R. Casazza PhD, RD/Assistant Professor, UAB, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F080605012
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: obesity, puberty, diabetes,insulin dynamics
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A, 1 (Experimental): low-carbohydrate (42%)
  Interventions: Other: Dietary
- A,2 (Experimental): standard carbohydrate (55%) based on ADA recommendations
  Interventions: Other: Dietary

INTERVENTIONS:
Other: Dietary — modification of macronutrient content

SUMMARY:
A diet (42% carbohydrate) specialized to the unique metabolic characteristics of peripubertal African AMerican girls (hyperinsulinemic, low insulin sensitive) will be more effective in maintaining glucose and insulin homeostasis compared to a standard diet (55% carbohydrate)

ELIGIBILITY:
Inclusion Criteria:

* African American girls aged 9-14,
* Overweight < 90th percentile

Exclusion Criteria:

* On medications known to affect metabolism prior disease diagnosis

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
decreased insulin secretion | 25 weeks

SECONDARY OUTCOMES:
decreased markers of inflammation; decreased estradiol concentration | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Krista Casazza, PhD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States